CLINICAL TRIAL: NCT00748449
Title: Acceptability and Effectiveness of Colonography Compared to Colonoscopy for the Detection of Advanced Adenomas in Patients at High Risk for Colorectal Cancer
Brief Title: Colonography Versus Colonoscopy in High Risk Patient
Acronym: COLO-TDM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No more inclusions
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P051074
Record Dates: First submitted 2008-07-31; First posted 2008-09-08 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-08

CONDITIONS: Colorectal Cancer
Keywords: Colorectal advanced adenoma; Colorectal cancer polypectomy (endoscopic); Colectomy; Colonoscopy with anaesthesia; CT-colonography
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): CT Colonography
  Interventions: Procedure: CT-colonography
- 2 (Active Comparator): Colonoscopy
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — 1 Colonoscopy
  Other Names: Colonoscopy or CT-colonography
  Arms: 2
Procedure: CT-colonography — 1 CT-colonography; Procedure/Surgery/Radiation
  Arms: 1

SUMMARY:
to evaluate the acceptability of CT-colonography compared to colonoscopy for the detection of advanced adenomas in subpopulations at high risk of colorectal.

DETAILED DESCRIPTION:
Secondary objective: to evaluate the medical and economic impact of the implementation of CT- colonography in this setting.Methodology: prospective multicenter randomized controlled trial with direct patient benefitN° of patients to be included: 600 Study follow-up :1 consultation and 3 phone contacts (M1, M6 and M12)Evaluation criteria:Main endpoint: acceptability of the colorectal cancer screening (% of enrolled patients having actually undergone the exploration)Secondary endpoints: - cost/effectiveness ratio of the 2 diagnostic tests with calculation of the economic and medical costs. - number of advanced adenoma detected in each group- number of CRC cases detected in each group

ELIGIBILITY:
Inclusion Criteria:

Surveillance of patients with a personal history of advanced adenoma or CRC:

* Informed consent obtained
* Age ≥ 18 and ≤ 80 years old
* History of advanced adenomatous polyps
* Or history of non metastatic CRC with curative surgery and without other treatment more than 2 years before enrollment.
* Previous medical examination

Screening of patients with a Family history of CRC at high risk:

* Informed consent obtained
* Age ≥ 18 and ≤ 80 years old
* First degree family history of colorectal cancer diagnosed <60yrs during the five previous years-Previous medical examination

Exclusion Criteria:

Personal histories

* Age < 18 or >80 years old
* history of non adenomatous polyps
* history of Metastatic CRC
* familial adenomatous polyposis, Peutz-Jeghers syndrome, hereditary non polyposis colorectal cancer (HNPCC), juvenile polyposis syndrome
* Familial history of familial adenomatous polyposis
* Personal history of subtotal colectomy (but not of hemicolectomy, to confer to inclusion criteria)
* Colonoscopy with a polyps resection dated more than 5 years and less than 2 years prior to enrollment.
* Enrollment in another protocol
* no health insurance affiliation Family histories
* Age < 18 or >80 years old
* Patients with one or several family histories of first degree colorectal cancer occured to unknown age or diagnosed after 60 years old.
* Eligible patients having already undergone colonoscopy screening
* no health insurance affiliation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who refuse to undergo an examination | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederic PRAT, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Cochin, Paris, France